CLINICAL TRIAL: NCT02335515
Title: Gastric Retention Time of Floating Gastro-Retentive Capsules in Male Healthy Subjects After Breakfast as Measured by Magnetic Resonance Imaging (MRI)
Brief Title: The Gastric Residence Time (GRT) of Soctec Capsule After a Standardized Breakfast
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SkyePharma AG (Industry)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SKY1049#10600-1-001
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Gastroretentive System; Gastric Retention Time (GRT); capsule; Soctec; Gastroenterology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Soctec / Capsule (Experimental): HS intakes one(1) Soctec Capsule after standardized breakfast
  Interventions: Device: Soctec

INTERVENTIONS:
Device: Soctec — Gastroretentive Drug Delivery System

SUMMARY:
The primary objective of the study was to assess the gastric residence time (GRT) of the Soctec capsule after a standardized breakfast. 12 healthy subjects will undergo an initial screening visit. Eligible subjects will undergo the study procedure. The hypothesis is that the GRT of the Soctect Capsule after a standardized breakfast and lunch will be longer compared to literature values reported for a simliar sized capsule.

ELIGIBILITY:
Inclusion Criteria:

* Male HS, aged between 18 and 50 years.
* Subjects must be in a good health and have BMI between 19 and 25 kg/m2.
* Subjects must be able to read, understand and sign the written informed consent.
* Subjects must be willing and able to comply with study requirements.

Exclusion Criteria:

* History of gastrointestinal, cardiorespiratory (including arterial hypertension), hematologic, renal, atopic, alimentary or psychiatric disorder, panic attacks, diabetes, drug or alcohol abuse.
* Subjects with a history of HIV, hepatitis B or hepatitis C.
* Requiring medication that might alter gut function, including anticholinergics, calcium channel blockers, beta blockers, laxatives, prokinetics, proton-pump inhibitors and non-steroidal anti-inflammatory drugs.
* Prior abdominal surgery other than uncomplicated appendectomy or hernia repair.
* Subject with claustrophobia (fear of small spaces).
* Presence of implants, devices or metallic foreign bodies that might interact with the MRI
* Participation in another investigational study where the study drug was received within 90 days prior to the screening visit.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
To assess the gastric residence time (GRT) of the Soctec Capsule after a standardized breakfast. | MRI scnas will be performed every 30 minutes starting after capsule intake for up to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Karim Bagate, PhD, Study Director — SkyePharma AG